CLINICAL TRIAL: NCT05984225
Title: Assessing the Impact of an Online Program Regarding Professional Ethics in Physiotherapy. A Prospective Clinical Trial
Brief Title: Impact of an Online Program in Ethics in Physiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, Assistant professor, PT, PhD, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BL_ETHICS_01
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Ethics, Narrative
Keywords: Learning; Ethics; Students; Knowledge; Physiotherapy
MeSH Terms: conditions — Narration

STUDY DESIGN:
Intervention Model Description: Interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapy students (Experimental): Physiotherapy students of the 2nd course of the Grade of Physiotherapy of the University of Valencia.
  Interventions: Other: Online learning

INTERVENTIONS:
Other: Online learning — The students performed a 10-week Online Learning (OL) program based on Professional Ethics. The program included:
  1. Synchronous learning (1 session/week, 1 hour each).
  2. Asynchronous learning: i) OL classes were recorded; ii) Moodle platform: for read breaking news, upload tasks or solve any doubt they may have through discussion forums; iii) An OL specific syllabus that consisted of five themes from the ethics knowledge; iv) An OL glossary, including the concept, explanation of the concept, and source; v) Bullet-point videos highlighting the most important issues of each theme; vi) Podcasts about Professional Ethics, Ethics in physiotherapy; vii) Links to websites; viii) Gamification using mobile Apps regarding ethical decision-making, healthcare, and Ethics or Professional Ethics, as well as an OL crossword; ix) OL activities were created and personalized comments about the activities were reported by the teachers to give feedback to the students.

SUMMARY:
Given the continuing ethical problems faced by physiotherapists, improving their students' ethical competence is relevant. The development of ethical decision-making skills is particularly important for students preparing to enter professional health careers like physiotherapy. According to the Bologna process, the education of physiotherapists includes the cultivation of relevant generic/transversal competencies, including ethical competence. To achieve this, diverse teaching, learning, assessment, and feedback strategies are necessary and helpful in facilitating the acquisition of these competencies.

The physiotherapist needs to carry out ethics efficiently through ethical reasoning and critical thinking to develop ethical decision-making abilities. Active learning methods allow us to get students to follow the highest ethical standards and successfully manage ethical situations in the workplace. Despite some studies showing physiotherapists have a deficit in clinical practice ethics.

However, there is a lack of research focusing on online learning (OL) physiotherapy ethics education, and studies of review on mixed health professionals many times do not include physiotherapy studies.

Considering this, the primary objective of this study is to assess the effectiveness of an OL program in developing ethical competence in physiotherapy students. Specifically, the study aims to evaluate the impact of the program on generic competences, knowledge acquisition, ethical sensitivity, engagement, and instructional design within the OL environment.

ELIGIBILITY:
Inclusion Criteria:

* To be studying the Physiotherapy Degree at the University of Valencia.

Exclusion Criteria:

* Not willing to participate.
* Students with previous ethics training.
* Not willing to provide the written consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Generic competencies | 0 week, 5 week, 10 week
  Questionnaire for the Evaluation of Generic Comeptences in Univesity Students. It is a 45-item instrument with a Likert scale from 1 = always to 6 = rarely, thus lower scores mean higher generic competencies. The internal consistency of this questionnaire is 0,92. Several competencies are assessed: 1) instrumental competencies (Job performance, Management skills); 2) systematic competencies (Leadership, Work motivation, Learning capabilities; 3) interpersonal competence (Interpersonal relationships and teamwork).

SECONDARY OUTCOMES:
Knowledge acquisition of Professional ethics | 0 week, 5 week, 10 week
  measured with a multiple-choice knowledge test. The test included fifteen multiple choice questions that assessed basic professional ethics concepts that physiotherapy students are required to know, such as moral values, ethics; bioethics and Professional Ethics in physiotherapy, ethical professional act, and legal professional act; professional ethical principles, physiotherapists deontological code, ethical situations, or professional values in physiotherapy. Students were not previously informed about retention exams to avoid any preparation for the test.
Ethical sensitivity | 0 week, 5 week, 10 week
  measured with the Ethical Sensitivity Scale Questionnaire (ESSQ). The ESSQ is based on Narvaez's theory of ethical sensitivity. The ESSQ is comprised of 28 items using a 4-point Likert scale (1 = totally disagree, 5 = totally agree), that are classified into seven dimensions: i) Reading and expressing emotions, ii) Taking the perspectives of others, iii) Caring by connecting to others, iv) Working with interpersonal and group differences, v) Preventing social bias, vi) Generating interpretations and options, vii) Identifying the consequences of actions and options. The higher score on the test is 5 points. A higher score showed greater ethical sensitivity. The reliability ranged between α = 0,63 (preventing social bias) and α = 0,79 (working with interpersonal and group differences). The overall reliability of this questionnaire is Cronbach's α = 0,81.
Engagement | Week 10
  with the Student Engagement Questionnaire. It is a 35-item questionnaire, scored on a five-point Likert scale (1 = totally disagree, 5 = totally agree). The questionnaire is divided into five dimensions: i) Intellectual capabilities (items 1-10); ii) Working together (items 11-16); iii), Teaching (items 17-25); iv) Teacher-student relationship (items 26-29); and v) Student-student Relationship (items 30-35). The maximum score of the questionnaire is 5 points. The higher the score, the higher the students´ engagement. Cronbach's α of this questionnaire ranges from 0.75 to 0.89.
Design of the Online Learning program instructions | Week 10
  using the Community of Inquiry Questionnaire. It is composed of 34 items scored on a five-point Likert scale (1 = strongly disagree, 5 = strongly agree) that includes three dimensions: i) Cognitive dimension (items 1-13), referring to the degree to which the participants are capable of construct meaning and knowledge through continuous communication, reflection, and discussion; ii) Social dimension (items 14-22), defined as the ability of the participants to identify with the community, communicate and develop interpersonal relationships; iii) Teaching dimension (items 23-34), referring to the design, guidance, and direction, by teachers, of cognitive and social processes to achieve significant learning results in students. The maximum score of the questionnaire is 5 points. Questionnaire validation shows satisfactory results (Cronbach's α being 0.90 for each dimension).

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, PT, PhD, Study Chair — University of Valencia
Locations (1):
- Faculty of Physiotherapy of the University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No